CLINICAL TRIAL: NCT04468061
Title: Saci-IO TNBC: Randomized Phase II Study of Sacituzumab Govitecan With or Without Pembrolizumab in PD-L1-negative Metastatic Triple Negative Breast Cancer (TNBC)
Brief Title: Sacituzumab Govitecan +/- Pembrolizumab in Metastatic TNBC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ana C Garrido-Castro, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-166
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; PD-L1 Negative
Keywords: Breast Cancer; Triple Negative Breast Cancer; PD-L1 Negative
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sacituzumab Govitecan + Pembrolizumab (Experimental): Participants will receive Sacituzumab Govitecan + Pembrolizumab at a pre-determined dose during a 21 day cycle.
  Sacituzumab Govitecan will be given on days 1 and 8 of the 21 day cycle Pembrolizumab will be given on day 1 of the 21 day cycle.
  Interventions: Drug: Sacituzumab Govitecan; Drug: Pembrolizumab
- Sacituzumab Govitecan (Experimental): Participants will receive Sacituzumab Govitecan at a pre-determined dose during a 21 day cycle.
  Sacituzumab Govitecan will be given on days 1 and 8 of a 21-day cycle
  Interventions: Drug: Sacituzumab Govitecan
- Retreatment (Experimental): Participants randomized to the combination arm (Sacituzumab Govitecan + Pembrolizumab) who stop with CR after at least 24 weeks of treatment may be eligible for additional pembrolizumab and/or sacituzumab govitecan therapy if they progress after stopping study treatment. This is termed the Second Course Phase and is only available if the study remains open and the subject meets conditions.
  .
  Interventions: Drug: Sacituzumab Govitecan; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Intravenous Infusion
  Other Names: IMMU-132; Trodelvy
Drug: Pembrolizumab — Intravenous Infusion
  Other Names: Keytruda
  Arms: Retreatment; Sacituzumab Govitecan + Pembrolizumab

SUMMARY:
This research study involves testing the safety and efficacy of an investigational intervention for patients with triple-negative breast cancer (TNBC) that has spread, or metastasized, to other parts the body and is PD-L1-negative.

The names of the study interventions involved in this study are:

* Sacituzumab govitecan (Trodelvy™;IMMU-132)
* Pembrolizumab (Keytruda®; MK-3475)

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug or a combination of investigational drugs to learn whether the drug or drug combination works in treating a specific disease. "Investigational" means that the drug or drug combination is being studied.

The U.S. Food and Drug Administration (FDA) has approved Sacituzumab Govitecan for metastatic triple-negative breast cancer, but it is currently approved only for patients who have had 2 or more prior regimens for metastatic disease. The U.S. Food and Drug Administration (FDA) has approved Pembrolizumab for metastatic triple-negative breast cancer, but it is currently approved only for patients with PD-L1-positive metastatic triple-negative breast cancer.

In this research study, we are:

* Studying Sacituzumab Govitecan alone or in combination with Pembrolizumab as a possible treatment for patients with metastatic triple-negative breast cancers that are PD-L1-negative.
* Sacituzumab Govitecan is composed of a chemotherapy drug, called Irinotecan, which is attached to an antibody. Antibodies are proteins normally made by the immune system that bind to substances that don't belong in the body to prevent harm. The antibody in this study binds to certain types of cancer tumors, including triple-negative breast tumors.
* Pembrolizumab is an immunotherapy, called an anti-PD-1 or a checkpoint inhibitor, and is an antibody (a type of human protein) designed to allow the body's own immune system to seek out and destroy tumors. It has been used in previous research studies to treat breast cancer, where it has been shown to be effective.
* The overall goal of this study is to evaluate the effectiveness of either Sacituzumab Govitecan alone or in combination with Pembrolizumab, in delaying the worsening of triple-negative breast cancers that are PD-L1-negative.

The research study procedures include: screening for eligibility, research blood collections, at least two research biopsies, paired research stool collections, questionnaires, data collection, and study treatment including evaluations and follow up visits.

Participants will be randomized into one of two groups.

* Group A: Sacituzumab Govitecan on days 1 and 8 and Pembrolizumab on day 1 of a 21-day cycle
* Group B: Sacituzumab Govitecan alone on days 1 and 8 of a 21-day cycle

Participants will receive study treatment for as long as they are benefitting from this therapy. Participants will be followed for the rest of their life.

It is expected that about 110 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer with unresectable locally advanced or metastatic disease. Participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* Estrogen-receptor and progesterone-receptor expression both ≤ 5% by immunohistochemistry (IHC), and HER2-negative status as determined by the current ASCO/CAP guidelines. If a patient has more than one histological result, the most recent sample will be considered for inclusion.
* Participants must have PD-L1-negative metastatic breast cancer defined as less than 1% expression of PD-L1 on tumor-infiltrating immune cells (IC) by the PD-L1 IHC SP142 assay or a Combined Positive Score (CPS) less than 10 by the PD-L1 IHC 22C3 assay measured with standard of care testing.
* Participants must be treatment-naïve in the metastatic setting.
* Participants must have evaluable or measurable disease per RECIST 1.1. Patients with bone only disease will be allowed to participate.
* Participants must agree to undergo a research biopsy, if tumor is safely accessible, at baseline. Previously collected archival tissue will also be obtained on all participants. Tissue needs to be located and availability confirmed at time of registration (see Section 9 for more details). Participants must agree to a mandatory repeat biopsy 3-6 weeks after starting treatment, if tumor is safely accessible.
* Prior chemotherapy: Participants must have received no prior chemotherapy for metastatic breast cancer and must have discontinued all chemotherapy at least 28 days prior to study treatment initiation. No prior irinotecan or topoisomerase I-containing antibody drug conjugates in the metastatic or neo/adjuvant setting are allowed. All toxicities related to prior chemotherapy must have resolved to CTCAE v5.0 grade 1 or lower, unless otherwise specified per protocol, except alopecia can be any grade and neuropathy can be grade 2 or lower.
* Prior biologic therapy: Patients must have received no prior biologic therapy for metastatic breast cancer and discontinued all biologic therapy at least 28 days prior to study treatment initiation. All toxicities related to prior biologic therapy must have resolved to CTCAE v5.0 grade 1 or lower, unless otherwise specified per protocol.
* Prior radiation therapy: Patients may have received prior radiation therapy. Radiation therapy must be completed at least 7 days prior to study treatment initiation, and all toxicities related to prior radiation therapy must have resolved to CTCAE v5.0 grade 1 or lower, unless otherwise specified per protocol. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
* Previously treated brain metastases are permitted, with the following provisions:

  * Prior SRS should complete ≥ 7 days before study treatment initiation
  * Prior WBRT should complete ≥ 7 days before study treatment initiation.
  * Any corticosteroid use for brain metastases must have been discontinued for ≥ 7 days prior to study treatment initiation.
* The subject is ≥ 18 years old.
* ECOG performance status 0-1 (Karnofsky > 60%, see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,000/mcL
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥ 9.0 g/dl
  * INR/PT/aPTT ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is in therapeutic range of anticoagulant
  * Total bilirubin ≤1.5 × institutional upper limit of normal (ULN)(or ≤2.0 x ULN in patients with documented Gilbert's Syndrome)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN or ≤5 × institutional ULN for participants with documented liver metastases
  * Serum creatinine ≤1.5 × institutional ULN OR creatinine clearance ≥ 30 mL/min/ 1.73m2 for participants with creatinine levels above institutional ULN.
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 2 weeks prior to study treatment initiation. Childbearing potential is defined as participants who have not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause) and have not undergone surgical sterilization (removal of ovaries and/or uterus).
* Women of childbearing potential (WOCBP) must agree to use an adequate method of contraception. Contraception is required starting with the first dose of study medication through 180 days (6 months) after the last dose of study medication. Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established and proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with pembrolizumab and 3 months after the last dose of study treatment
* Participants on bisphosphonates or RANK ligand inhibitors may continue receiving therapy during study treatment and also may initiate therapy with these agents on study if clinically indicated.
* The participant must be capable of understanding and complying with the protocol and willing to sign a written informed consent document.

Exclusion Criteria:

* Has received prior systemic anti-cancer therapy, including investigational agents, within 4 weeks of study treatment initiation or during the course of this study (bisphosphonates and RANK ligand inhibitors are allowed).
* Prior therapy with any anti-PD-1, PD-L1, or PD-L2 agent or sacituzumab govitecan (IMMU-132). Prior therapy with irinotecan or topoisomerase I-containing antibody drug conjugates at any time for early stage or metastatic disease.
* Prior hypersensitivity to pembrolizumab or the excipients of pembrolizumab or sacituzumab govitecan (IMMU-132 therapy).
* Known history of UDP-glucuronosyltransferase 1A1 (UGT1A1) *28 allele homozygosity, which is associated with increased risk for neutropenia and diarrhea related to irinotecan. Note: Concurrent administration of strong UGT1A1 inhibitors or inducers is not allowed during the course of the study.
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms.
* Major surgery within 2 weeks prior to study treatment initiation. Patients must have recovered from any effects of any major surgery.
* Uncontrolled, significant intercurrent or recent illness including, but not limited to, ongoing or active infection, uncontrolled non-malignant systemic disease, uncontrolled seizures, or psychiatric illness/social situation that would limit compliance with study requirements in the opinion of the treating investigator.
* Participant has a medical condition that requires chronic systemic steroid therapy (> 10 mg of prednisone daily or equivalent) or any other form of immunosuppressive medication (including disease modifying agents) and has required such therapy in the last 2 years. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic therapy.
* Participant has documented history of autoimmune disease or syndrome that currently requires systemic steroids or immunosuppressive agents.
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Individuals with a history of a second malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers that have been diagnosed and treated within the past 3 years are eligible: cervical/prostate carcinoma in situ, superficial bladder cancer, non-melanoma cancer of the skin. Patients with other cancers diagnosed within the past 3 years and felt to be at low risk of recurrence should be discussed with the study principal investigator to determine eligibility.
* Participant has a known history of human immunodeficiency virus (HIV), Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as detected HCV RNA [qualitative]) infection. HIV-positive participants are ineligible due to the potential for pharmacokinetic interactions of combination antiretroviral therapy with study drugs and the increased risk of fatal infections when treated with marrow-suppressive therapy. Note: No testing for HIV, Hepatitis B, or Hepatitis C is required unless mandated by local health authority.
* The participant has received a live vaccine within 28 days prior to study treatment initiation. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine. The use of the inactivated seasonal influenza vaccine is allowed.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* It is unknown whether pembrolizumab is excreted in human milk. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant, participants who are breast-feeding are not eligible for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 3 years
  Compare PFS of patients randomized to receive sacituzumab govitecan in combination with pembrolizumab (Arm A) versus those randomized to receive sacituzumab govitecan monotherapy (Arm B).
  Defined as the time from study randomization to disease progression, per RECIST 1.1 or medical judgment, the latter based on established clinical parameters, such as rising tumor markers and physical exam evidence of progression, i.e. worsening chest wall disease, or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing Overall Survival (OS), defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive, will be reported with Kaplan Meier estimates.
Objective Response Rate (ORR) | 3 years
  Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing Objective Response Rate by RECIST 1.1.
Duration of response (DOR) | 3 years
  Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing the duration of response (the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented or death due to any cause. Participants without events reported are censored at the last disease evaluation).
Time to objective response (TTOR) | 3 years
  Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing the time to objective response defined as the time from randomization to the date of the first documented CR or PR (whichever is first recorded).
Time to progression (TTP) | 3 years
  Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing Time to progression (TTP) defined as the time from randomization (or registration) to progression, or censored at date of last disease evaluation for those without progression reported.
Clinical benefit rate (CBR) | 3 years
  Compare the efficacy of sacituzumab govitecan with pembrolizumab to that of sacituzumab govitecan alone by assessing Clinical benefit rate (CBR) according to RECIST 1.1, defined as CR, PR or stable disease for ≥ 24 weeks.
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | 3 years
  Evaluate the safety and tolerability of sacituzumab govitecan and pembrolizumab compared to sacituzumab govitecan alone by monitoring adverse events, including immune-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Ana C Garrido-Castro, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (14):
- United States (14):
  - Stamford Hospital, Stamford, Connecticut
  - Miami Cancer Institute at Baptist Health (Kendall), Miami, Florida
  - Miami Cancer Institute at Baptist Health, Plantation, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Eastern Maine Medical Center, Brewer, Maine
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - DFCI @ Foxborough, Foxborough, Massachusetts
  - DFCI @ Milford Regional Hospital, Milford, Massachusetts
  - DF/BWCC in Clinical Affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pennsylvania-Abramson Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research Institute, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: https://www.dana-farber.org/research/innovations

REFERENCES:
- [Derived] Kwapisz D. Sacituzumab Govitecan-hziy in Breast Cancer. Am J Clin Oncol. 2022 Jul 1;45(7):279-285. doi: 10.1097/COC.0000000000000919. Epub 2022 May 12. PMID 35728046